CLINICAL TRIAL: NCT04542863
Title: The Molecular Imaging Research of F-18 Labeled DX600 PET Probe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020KT102
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging cohort (Experimental): All study participants will be allocated to this arm (single-arm study). Study participants will undergo 18F-DX600 PET/CT scans.
  Interventions: Other: 18F-DX600 PET/CT

INTERVENTIONS:
Other: 18F-DX600 PET/CT — DX600, labeled with 18F will be used as a molecular imaging tracer for PET/CT scanning

SUMMARY:
Angiotensin-converting enzyme 2 (ACE2) plays an important role in renin-angiotensin system (RAS) and has been reported to relate with cancer. Recently, it has also been proved as the key target for COVID-19 infection.

DX600 is a polypeptide that can specific binding to ACE2 specifically with nanomolar affinity reported in literature. This study constrcuted a radio-tracer, DX600 Labeled by PET Radionuclide, to monitoring biodistribution ACE2 in human beings, evaluate the detection ability of radio-tracer in ACE2 over-expression tumors and dynamic changes of ACE2 expression under therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >3 years old; both sex;
* ECoG 0 or 1;
* Patients that would undergo biopsy or surgical operation with high ACE2 expression tumors such as colorectal cancer, renal cancer, pancreatic cancer, gastric cancer, liver cancer, lung cancer, brain cancer or suspected tumor.
* use 18F-FDG PET/CT as baseline evaluation

Exclusion Criteria:

* Significant hepatic or renal dysfunction;
* Is Pregnant or ready to pregnant;
* Cannot lie on their back for half an hour;
* Suffering from claustrophobia or other mental diseases;
* Refusal to join the clinical study;

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value (SUV) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No